CLINICAL TRIAL: NCT02392572
Title: Phase I/II Study of Oral ONC201 in Patients With Relapsed or Refractory Acute Leukemias and High-Risk Myelodysplastic Syndromes
Brief Title: ONC201 in Treating Patients With Relapsed or Refractory Acute Leukemia or High-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0731; NCI-2015-00504 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20152152; 1-907936-1; 1159166; 1-910469-1; 204710; 2014-0731 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — TIC10 compound; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Akt/ERK inhibitor ONC201) (Experimental): Patients receive Akt/ERK inhibitor ONC201 PO once every 3 weeks. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Drug: Venetoclax
- Arm B (Akt/ERK inhibitor ONC201) (Experimental): Patients receive Akt/ERK inhibitor ONC201 PO once every week. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Drug: Venetoclax
- Arm C (Akt/ERK inhibitor ONC201) (Experimental): Patients receive Akt/ERK inhibitor ONC201 PO on the first two consecutive days of every week. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Drug: Venetoclax
- Arm D (Akt/ERK inhibitor ONC201) (Experimental): Patients receive Akt/ERK inhibitor ONC201 PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Drug: Venetoclax
- Arm E (Akt/ERK inhibitor ONC201) (Experimental): Arm E (Akt/ERK inhibitor ONC201) Patients receive Akt/ERK inhibitor ONC201 PO twice weekly for 4 weeks and venetoclax daily on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Drug: Venetoclax

INTERVENTIONS:
Drug: Akt/ERK Inhibitor ONC201 — Given PO
  Other Names: ONC-201; ONC201; TIC10
Drug: Venetoclax — Given PO
  Other Names: Venclexta; ABT-199; GDC-0199

SUMMARY:
This phase I/II trial studies the side effects and best dose of ONC201 and to see how well it works in treating patients with acute leukemia or high-risk myelodysplastic syndrome that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). ONC201 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine recommended phase II dose for oral ONC201 ([Akt/ERK inhibitor ONC201) alone or in combination with VENETOCLAX in patients with relapsed or refractory acute myelogenous leukemia (AML), myelodysplastic syndrome (MDS) or acute lymphoblastic leukemia (ALL). (Phase I) II. To identify toxicities associated with oral ONC201 alone or in combination with VENETOCLAX in patients with relapsed or refractory AML, MDS or ALL. (Phase I) III. To determine the objective response rate to ONC201 alone in patients with relapsed or refractory AML, MDS or ALL. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics (PK) of oral ONC201 alone or in combination with VENETOCLAX. (Phase I) II.To observe the anti-tumor effects of oral ONC201 alone or in combination with VENETOCLAX in patients with relapsed or refractory AML, MDS or ALL. (Phase I) III. Confirm tolerability of recommended phase II dose. (Phase II) IV. Assess clinical outcomes associated with ONC201 alone or in combination with VENETOCLAX in patients with relapsed or refractory AML, MDS or ALL. (Phase II) V. Correlate clinical outcome with tumor and serum biomarkers. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study. Patients are assigned to 1 of 5 arms.

ARM A: Patients receive Akt/ERK inhibitor ONC201 orally (PO) once every 3 weeks. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive Akt/ERK inhibitor ONC201 PO once every week. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive Akt/ERK inhibitor ONC201 PO on the first two consecutive days of every week. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive Akt/ERK inhibitor ONC201 PO once daily (QD). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive Akt/ERK inhibitor ONC201 PO twice weekly. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM F: Patients receive Akt/ERK inhibitor ONC201 PO twice weekly for 4 weeks and venetoclax daily on days 1-21 every 28 day cycle.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* For Arms A, B, C, D, E, F patients must have relapsed or refractory acute leukemias or high-risk MDS for which no standard therapies are anticipated to result in a durable remission
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device, such as a condom, diaphragm, or cervical/vault cap), for 16 weeks after the last dose of study drug, and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial; nursing patients are excluded; sexually active men must also use acceptable contraceptive methods for the duration of time on study and for at least 16 weeks after the last dose of study drug; pregnant and nursing patients are excluded because the effects of ONC201on a fetus or nursing child are unknown
* Must be able and willing to give written informed consent
* The interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents or at least 5 half-lives for noncytotoxic agents; if the patient is on hydroxyurea to control peripheral blood leukemic cell counts, the patient must be off hydroxyurea for at least 24 hours before initiation of treatment on this protocol; persistent clinically significant toxicities from prior therapy must not be greater than grade 1
* Serum creatinine < 2.0 mg/dl
* Total bilirubin =< 1.5 x the upper limit of normal (ULN) unless considered due to Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 3 x the ULN unless considered due to organ leukemic involvement
* Relapse > 6 months since autologous or allogeneic stem cell transplantation provided:

  * No active graft-versus-host disease (GVHD > grade 1)
  * No treatment with high dose steroids for GVHD (up to >= 20 mg prednisolone or equivalent per day)
  * No treatment with immunosuppressive drugs with the exception of low dose cyclosporine and tacrolimus

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure (New York Heart Association class III and IV), uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure (New York Heart Association class III and IV)
* Patients receiving any other standard or investigational treatment for their hematologic malignancy within past 2 weeks for cytotoxic agents or at least 5 half-lives for noncytotoxic agents
* Subject has been diagnosed or treated for another malignancy within 3 years of enrolment, except in situ malignancy, or low-risk prostate, skin or cervix cancer after curative therapy
* Known history of seropositive for human immunodeficiency virus (HIV) antibodies (HIV1 and HIV2), hepatitis C antibody (Hep C Ab) or a hepatitis B carrier (positive for hepatitis B surface antigen [HBsAg])
* Active drug use or alcoholism
* Known or active central nervous system (CNS) involvement by leukemia
* White blood cell count more than 25 x 109/L prior to initiation of venetoclax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ONOC201 in Relapsed or Refractory Acute Myelogenous Leukemia (AML), Myelodysplastic Syndrome (MDS) or Acute Lymphoblastic Leukemia (ALL) | 21 days
  MTD is defined as the highest dose level in which 6 patients have been treated with at most 1 instance of dose limiting toxicity (DLT). Toxicities defined according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. DLT defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications and occurring during the first cycle on study that meets any of the following criteria:
  CTCAE grade 3 AST (SGOT) or ALT (SGPT) for > 7 days CTCAE grade 4 AST (SGOT) or ALT (SGPT) of any duration All other clinically significant NCI common terminology criteria that are CTCAE grade 3 or 4 (except for electrolyte disturbances responsive to correction within 24 h, diarrhea, nausea and vomiting that responds to standard medical care)
Objective Response (OR) (Phase II) | 63 days
  Objective responses for patients with AML and ALL include Complete Remission (CR), Complete Remission with Incomplete Blood Count Recovery (CRi), Partial Remission (PR) and morphologic leukemia-free state(Cheson and others, 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT02392572/ICF_000.pdf